CLINICAL TRIAL: NCT06946433
Title: Ensayo clínico Fase 1 de tDCS en Adultos Con TEA y/o TDAH Sin Discapacidad Intelectual
Brief Title: tDCS in Adults With ASD and/or ADHD Without Intellectual Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR (AG) 218_2022
Record Dates: First submitted 2025-04-08; First posted 2025-04-27 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder; Attention Deficit Disorder With Hyperactivity
Keywords: tdcs; autism; adhd
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Autistic Disorder | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active tDCS + Cognitive Training (Active Comparator): Participants in this arm will receive anodal transcranial direct current stimulation (tDCS) at 2 mA for 20 minutes per session over 10 consecutive workdays. The anode will be placed over the left dorsolateral prefrontal cortex (F3) and the cathode over the right frontopolar cortex (Fp2) using the 10-20 EEG system. Stimulation will be administered concurrently with cognitive training using the NeuronUP platform, which includes tasks targeting attention, memory, and executive function.
  Interventions: Device: Transcranial Direct Current Stimulation - Active; Behavioral: Cognitive Training
- Sham tDCS + Cognitive Training (Sham Comparator): Participants in this arm will undergo the same setup and procedures as the active tDCS group but will receive sham stimulation, which mimics the sensation of tDCS without delivering current beyond the initial ramp-up/down. They will also complete cognitive training with the NeuronUP platform during each session.
  Interventions: Device: Transcranial Direct Current Stimulation - Sham; Behavioral: Cognitive Training

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation - Active — This intervention involves non-invasive brain stimulation using transcranial direct current stimulation (tDCS) delivered via saline-soaked sponge electrodes. The anode is placed at F3 (left dorsolateral prefrontal cortex) and the cathode at Fp2 (right frontopolar cortex), according to the international 10-20 EEG system. A 2 mA current is applied for 20 minutes per session, administered once daily on 10 consecutive workdays.
  During stimulation, participants engage in cognitive training using the NeuronUP platform, which provides structured, interactive tasks designed to train executive function, attention, and working memory. This combination aims to enhance neural plasticity by pairing neuromodulation with cognitive engagement.
  Arms: Active tDCS + Cognitive Training
Device: Transcranial Direct Current Stimulation - Sham — The sham condition mimics the active setup but delivers only brief ramp-up/down stimulation, producing the initial sensation without sustained current.
  Arms: Sham tDCS + Cognitive Training
Behavioral: Cognitive Training — The cognitive training intervention in this study is delivered through NeuronUP, a digital platform offering evidence-based cognitive stimulation activities. This intervention targets core cognitive domains such as working memory, attention, and executive function through personalized, interactive tasks. What distinguishes this approach is NeuronUP's extensive library of over 10,000 activities, its ability to tailor difficulty levels in real time based on individual performance, and the inclusion of functional tasks that mirror real-life scenarios. Unlike other interventions, NeuronUP also enables therapist-guided customization, allowing for individualized treatment plans that evolve with participant progress, ensuring both relevance and ecological validity.

SUMMARY:
The goal of this clinical trial is to learn about the safety and tolerability of transcranial direct current stimulation (tDCS) combined with cognitive training in adults with Autism Spectrum Disorder (ASD) and/or Attention-Deficit/Hyperactivity Disorder (ADHD).

The main question it aims to answer is:

Is tDCS safe and well-tolerated in adults with ASD and/or ADHD?

Researchers will compare active tDCS to a sham (placebo-like) stimulation to evaluate safety and tolerability.

Participants will:

Receive either active or sham tDCS for 20 minutes daily over 10 consecutive workdays

Undergo stimulation with the anode placed at F3 and the cathode at Fp2

Complete daily cognitive training exercises using the NeuronUP platform during stimulation

Attend baseline and follow-up assessments to monitor for any side effects or discomfort related to the intervention

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 to 55 years

Clinical diagnosis of Autism Spectrum Disorder (ASD) and/or Attention-Deficit/Hyperactivity Disorder (ADHD) confirmed via medical records or structured clinical interview

Able to provide informed consent

Fluent in the language used for assessments and cognitive training tasks

Stable medication regimen (if applicable) for at least 4 weeks prior to enrollment

Willing and able to attend 10 consecutive weekday sessions and follow-up assessment

Exclusion Criteria:

History of epilepsy, seizures, or significant neurological disorder (e.g., traumatic brain injury, stroke)

Current diagnosis of psychotic disorder or bipolar disorder

Presence of metal implants in the head (excluding dental work), pacemaker, or other contraindications to tDCS

Current substance use disorder (within past 6 months)

Pregnant or planning to become pregnant during the study period

Participation in another intervention study within the last 30 days

Any condition that, in the opinion of the investigators, may make participation unsafe or interfere with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Throughout the 10-day intervention period and at follow-up (up to 2 weeks post-intervention)
  Participants will be monitored for adverse events, side effects (e.g., headache, skin irritation, fatigue), and dropout rates. This will be assessed through participant self-report, clinician observation, and standardized side effect checklists administered during and after each session. The outcome will help determine whether daily tDCS paired with cognitive training is safe and acceptable for adults with ASD and/or ADHD.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No